CLINICAL TRIAL: NCT02602795
Title: Distress Tolerance and HIV Prevention With XR-NTX Initiation in Opioid Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34DA037797 (NIH)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2017-04

CONDITIONS: Opiate Dependence; Sexually Transmitted Diseases; HIV
Keywords: Opiate Dependence; Sexually Transmitted Diseases; HIV; Extended release naltrexone
MeSH Terms: conditions — Opioid-Related Disorders; Sexually Transmitted Diseases | interventions — Acceptance and Commitment Therapy; Information Motivation Behavioral Skills Model

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Distress Tolerance (DT) (Experimental): Acceptance and Commitment Therapy based Distress Tolerance (DT) intervention to facilitate opioid detoxification delivered in six 50-minute individual telehealth sessions.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- HIV/STI Intervention (Active Comparator): Information Motivation Behavioral model based HIV/STI risk reduction intervention delivered in six 50-minute individual telehealth sessions.
  Interventions: Behavioral: Information Motivation Behavioral Model
- Treatment As Usual (TAU) (No Intervention): Traditional treatment given to patients who elect to transition to XR-NTX at the treatment sites.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The intervention is based on Acceptance and Commitment Therapy and will be tailored to help participants develop target adaptive responses to negative affect and other negative internal stimuli related to opioid detoxification.
  Arms: Distress Tolerance (DT)
Behavioral: Information Motivation Behavioral Model — This intervention is based on the Information Motivation Behavior model for HIV/STI risk reduction and is tailored to more directly address HIV/STI risk among opioid dependent patients.
  Arms: HIV/STI Intervention

SUMMARY:
Before starting treatment with XR-NTX, a medication that blocks the positive effects of opioids and helps people stay off opioids, individuals who are dependent on opioids first have to endure a difficult withdrawal process. This study aims to develop and test an intervention to help people who are opioid dependent successfully complete that transition; the investigators will also develop and test a comparison condition aimed at reducing HIV risk behavior.

DETAILED DESCRIPTION:
Opioid dependence is a serious and increasingly pervasive problem. Opioid dependent individuals are at significantly increased risk for a wide range of physical and psychological problems including HIV and STIs. Extended-release naltrexone (XR-NTX) is an effective treatment for opioid dependence, but it requires that opioid-dependent individuals be completely opioid-free prior to its initiation to avoid precipitated withdrawal. The great majority of individuals attempting to cease opioid use will relapse before initiation of XR-NTX because of opioid withdrawal symptoms during detoxification. Distress Tolerance (DT) focused psychosocial interventions are well suited to address the clinical phenomena experienced by individuals withdrawing from opioids.

The purpose of this project is to develop a DT intervention to improve detoxification outcomes and an active comparison intervention targeting HIV and STI (HIV/STI) risk behavior. The DT intervention will be adapted from Acceptance and Commitment Therapy (ACT). The HIV/STI risk behavior intervention will target behaviors that put patients at risk for HIV and STIs including unprotected sex and needle sharing, as well as promoting regular HIV testing. Both interventions will be delivered through a telehealth videoconferencing system. If the HIV/STI intervention is found to result in reduced HIV/STI risk behavior and more frequent HIV testing, relative to the DT intervention, the investigators will incorporate its components into the DT intervention prior to launching a large-scale clinical trial. The long-term objective of this research program is to improve substance use and HIV/STI outcomes for opioid dependent individuals attempting to cease opioid use.

In Phase 1 of this project, the investigators will develop and pilot a DT intervention for individuals transitioning to XR-NTX and a time-matched HIV/STI risk reduction comparison intervention; both will be developed using an iterative process of piloting and modification based on data collected from pilot participants. In Phase 2, opioid dependent individuals transitioning to XR-NTX will be randomly assigned to DT, HIV/STI, or Treatment-As-Usual. All patients will receive medication assisted detoxification from the study recruitment site. It is expected that, as a result of this project, the investigators will have developed a well-specified and novel DT intervention tailored to meet the needs of opioid dependent patients transitioning to XR-NTX, the efficacy of which can be further tested in future Stage II randomized controlled trials. If found to be efficacious, this intervention will serve as an effective means of facilitating detoxification and opioid antagonist initiation, reducing the individual and societal burden due to opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

* Must (1) meet Diagnostic and Statistical Manual of Mental Disorders-IV Lifetime criteria for Opioid Dependence, (2) not plan to receive opioid agonist treatment or opioid analgesics, (3) have no medical need for opioid pain medication, (4) have Alanine Transaminase and Aspartate Aminotransferase < 150, and (5) have platelets > 90.

Exclusion Criteria:

* Must not (1) be currently psychotic, (2) have current drug or alcohol dependence that requires medical detoxification or a higher level of care that would interfere with study participation, (3) be pregnant or lactating, (4) have acute hepatitis or liver failure, (5) have a bleeding disorder, or (6) be allergic to XR-NTX components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Successful Detoxification | 6-months
  The investigators will compare the odds of successful detoxification, or receipt of the first XR-NTX injection, between treatment groups.
Number of XR-NTX Injections Received | 6-months
  The treatment groups will be compared on the number of XR-NTX injections received during follow-up.
Opioid Drug Use Outcomes | 6-months
  Percent of opioid use days compared between the groups
Illicit Drug Use Outcomes | 6-months
  Percent of illicit drug use days compared between the groups

SECONDARY OUTCOMES:
Sex Risk Behavior | 6-months
  The investigators will compare the occurrence of sex risk behavior between the treatment groups.
Drug Risk Behavior | 6-months
  The investigators will compare the occurrence of drug risk behavior between the treatment groups.
HIV Risk Behavior | 6-months
  The investigators will compare the occurrence of overall HIV risk behavior between the treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Ramsey, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States